CLINICAL TRIAL: NCT01845727
Title: Safety, Pharmacokinetics, and Efficacy of Topical 3% Amphotericin B Cream for the Treatment of Uncomplicated Cutaneous Leishmaniasis in Colombia
Brief Title: Topical 3% Amphotericin B Cream for the Treatment of Cutaneous Leishmaniasis in Colombia
Acronym: Anfoleish
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Drugs for Neglected Diseases (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DNDi-CL-TF001
Record Dates: First submitted 2013-04-24; First posted 2013-05-03 (Estimated); Last update posted 2016-07-26 (Estimated); Status verified 2016-07

CONDITIONS: Cutaneous Leishmaniasis
Keywords: Cutaneous leishmaniasis; Topical treatment; Colombia
MeSH Terms: conditions — Leishmaniasis, Cutaneous

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Topical Amphotericin B three times per day (Experimental): Anfoleish applied 3 times per day for 4 weeks (TID group)
  Interventions: Drug: Topical Amphotericin B at 3%
- Topical Amphotericin B two times per day (Experimental): Anfoleish applied 2 times per day for 4 weeks (BID group)
  Interventions: Drug: Topical Amphotericin B at 3%

INTERVENTIONS:
Drug: Topical Amphotericin B at 3%
  Other Names: Anfoleish

SUMMARY:
The proposed study encompasses a two-step approach. The first aiming to determine the safety of Topical 3% Amphotericin B Cream when applied three or two times per day for 4 weeks in subjects with un-complicated Cutaneous leishmaniasis (CL) whilst the second focusing in having and indication of the efficacy of the two above mentioned regimens of Topical 3% Amphotericin B Cream

For the first step, 30 subjects will be randomly assigned to receive direct observed treatment (DOT) with Topical 3% Amphotericin B Cream applied either three or two times per day for 4 weeks. Enrolment will be temporarily halted until all 30 subjects (15 in each group) have been enrolled and completed the 28 day treatment course. An interim analysis of all safety (Adverse Events, including local reactions and lab parameters) and pharmacokinetics collected on subjects who were randomized will be performed by data safety monitoring board. If no serious adverse events (SAEs) related to the study drug are identified on the first 30 subjects by the end of the treatment course, 50 additional subjects will be randomly allocated to receive Topical 3% Amphotericin B Cream either three or two times per day for 28 days

Subjects will have a follow-up visit at the end of therapy, on Day 45± 5 days, Day 63± 5 days and on Days 90± 14 days and on Day 180, minus 14d, plus 4 weeks to assess efficacy, as measured by the number of subjects who fulfil the cure criteria: 100% re-epithelialization of the lesion(s) by Day 90 and no relapse by Day 180. All subjects will be followed up to Day 180 for final analysis of efficacy.

ELIGIBILITY:
Inclusion Criteria:

* Subject with a confirmed infection due to L. braziliensis by polymerase chain reaction assay
* Subject has a lesion that satisfies the following criteria:
* ulcerative in character
* ulcer size equal or more than 0.5 cm and 3 cm (Longest diameter)
* not located on the ear, face, close to mucosal membranes, joints or on a location that in the opinion of the PI is difficult to maintain application of study drug topically.
* Subject with up to 3 lesions.
* Duration of lesion less than 3 months by patient history
* Subject able to give written informed consent and that the opinion of the investigator, the subject is capable of understanding and complying with the protocol

Exclusion Criteria:

* Female with a positive serum pregnancy test at screening or who is breast feeding, lactating or female at fertile age who does not agree to take appropriate contraception during treatment period up to Day 45.
* History of clinically significant medical problems or treatment that might interact, either negatively or positively, with topical treatment of leishmaniasis including any immunocompromising condition.
* Within 8 weeks (56 days) of starting study treatments, received treatment for leishmaniasis with any medication including antimonials likely, in the opinion of the PI, to modify the course of the Leishmania infection
* Has diagnosis or suspected diagnosis of mucocutaneous leishmaniasis based on physical exam.
* History of known or suspected hypersensitivity or idiosyncratic reactions to amphotericin
* Has laboratory values at screening as follow: Haemoglobin below 10 grams, Serum creatinine above normal level, alanine aminotransferase and or aspartate aminotransferase 3 times above normal range

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2014-02; Primary Completion 2016-05 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Proportion and severity of local adverse events of Anfoleish or Vehicle when applied three or two times per day. | At the end of treatment (Day 28)
  Local adverse events including erythema/redness, swelling/oedema, and vesicles will be scored according the following criteria:
  Grade 1: Visibly present but not associated with any other symptoms. Grade 2: Visibly present, large area around lesion site, and associated with other symptoms such as itching or pain. Medical intervention may be required.
  Grade 3: Severe symptoms that require medical discontinuation of the study drug.
Clinical cure rates in two regimens of Anfoleish: Three times a day and Two times a day | Day 90
  Cure is defined as 100% re-epithelialization of the lesion(s) by Day 90.

SECONDARY OUTCOMES:
Determination of Amphotericin B Cmax and Tmax in subjects treated with Anfoleish three or two times per day. | Day 45
Proportion and severity of laboratory adverse events of Anfoleish or vehicle when applied three or two times per day | At the end of treatment (Day 28
  Laboratory adverse events are limited to monitoring serum levels of creatinine, alanine aminotransferase and aspartate aminotransferase.

OTHER OUTCOMES:
Proportion of subjects showing a lesion's relapse by Day 180 | Day 180
  Relapse defined as a lesion that achieved 100% re-epithelialization by Day 90 that subsequently reopened by Day 180.

CONTACTS AND LOCATIONS:
Overall Officials: Ivan Dario Velez, Prof, Principal Investigator — PECET, Universidad de Antioquia, Medellin, Colombia
Locations (1):
- Programa de Estudios y Control de Enfermedades Tropicales (PECET), Universidad de Antioquia, Medellín, Colombia

REFERENCES:
- [Derived] Lopez L, Velez I, Asela C, Cruz C, Alves F, Robledo S, Arana B. A phase II study to evaluate the safety and efficacy of topical 3% amphotericin B cream (Anfoleish) for the treatment of uncomplicated cutaneous leishmaniasis in Colombia. PLoS Negl Trop Dis. 2018 Jul 25;12(7):e0006653. doi: 10.1371/journal.pntd.0006653. eCollection 2018 Jul. PMID 30044792